CLINICAL TRIAL: NCT03026270
Title: Effect of Therapeutical Paraffin Wax Bath in the Malleability of Burned Skin
Brief Title: Effect of Therapeutical Paraffin in the Malleability of Burned Skin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Elaine Caldeira de Oliveira Guirro, Professor Doctor postgraduation Program in Rehabilitation and Functional Performance, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 13386/2011
Record Dates: First submitted 2016-11-19; First posted 2017-01-20 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Burn
Keywords: Physiotherapy; Paraffin; Burn; Contracture
MeSH Terms: conditions — Burns; Contracture | interventions — Paraffin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- seven layers (Other): Volunteers will be submitted to the application of seven layers therapy paraffin surrounded by a plastic film film remaining in the area for 15 minutes, and then discarded. .The Application will be made with the patient in the supine position at rest for at least 10 min, then with an appropriate brush (5 cm wide)
  Interventions: Other: Paraffin
- ten layers (Other): Volunteers will be submitted to the application of seven layers therapy paraffin surrounded by a plastic film film remaining in the area for 15 minutes, and then discarded. .The Application will be made with the patient in the supine position at rest for at least 10 min, then with an appropriate brush (5 cm wide)
  Interventions: Other: Paraffin

INTERVENTIONS:
Other: Paraffin — The application of paraffin wax will be performed with the patient in the supine position at rest for at least 10 min, then with an appropriate brush (5 cm wide), will spend several layers with the brush into two distinct groups, seven or ten layers depending on the outcome of randomisation, in the region of interest of the upper limb, being scarred, surrounded by a plastic film film remaining in the area for 15 minutes, and then discarded

SUMMARY:
Effect of therapeutical paraffin wax bath in the malleability of burned skin

DETAILED DESCRIPTION:
The altered biomechanical properties of the skin entail limitation of movement, it have been important the statement of resources aimed at increasing skin suppleness. The objective of the study is to evaluate the effect of therapeutic paraffin in biophysical characteristics of the burned skin with or without scar hypertrophic. For this, 60 volunteers will be evaluated in the age group of 18-60 years, of both sexes, with deep second degree and third degree burns and evaluated areas submitted to therapeutic procedures, divided evenly into scar areas and normal skin. Applications will be set randomly by lot, with cross design (cross-over), and a minimum interval of seven days (wash-out) of the activities. The biophysical and biomechanical parameters of the skin will be assessed noninvasively by Cutometer of the model (MPA) 580, device to measure elasticity of the upper skin layer using negative pressure, and the durometer, measure hardness of the skin, before, immediately after 0, 10, 20 and 30 minutes of intervention with therapeutic paraffin in different procedures (number of layers and thermal insulation). Sociodemographic, clinical and surgical data of the volunteers will be evaluated by SPSS 15 (Statistical Analysis Software). The normality of the data will be verified by the Shapiro-Wilk test, and the effect of therapeutic procedures over time evaluated by the Friedman test (intragroup) and the test Kruskal-Wallis post hoc Dunn for comparisons between different funds (intergroup), p <0.05, will evaluated by software SPSS.

ELIGIBILITY:
Inclusion Criteria:

* Will be included in the study individuals who were victims of 2 deep burns or 3rd grade being subjected to grafting autogenous procedures, with or without the presence of hypertrophic scar, normal skin of individuals, ie without tissue damage and to agree to sign the term free and informed consent.

Exclusion Criteria:

* They will be included in this study individuals with diseases or deformities that affect the structure and function of the skin.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Distensibility of burned hypertrophic scar | up to 30 minutes
  Will be evaluated through the Cutometer®-MPA 580 of the intervention with therapeutic paraffin, being constituted by a small probe with diameter of 4 mm coupled in the equipment. The mechanism of action consists of deformation of the skin caused by suction, ie negative pressure giving a measured value. Once applied to the skin, an infrared light and a sensor located inside the probe perform the measurement of the distension of the skin during the period of continuous suction, followed by the phase of off where there is no suction.

SECONDARY OUTCOMES:
Hardness of burned hypertrophic scar before, immediately after 0, 10, 20 and 30 minutes. | up to 30 minutes
  The instrument was used immediately after 0, 10, 20 and 30 minutes of therapeutic paraffin intervention, always in a position perpendicular to the surface of the skin to minimize errors due to the inclination of the device and repeated three times , To obtain an average of values, intervals for 10 seconds between evaluations (Klinger, et al., 2013)

IPD SHARING:
Plan to Share IPD: Undecided